CLINICAL TRIAL: NCT02857192
Title: Study of Phenotypic and Functional Characteristics of Regulatory T Lymphocytes in Giant Cell Arteritis (Horton's Disease)
Brief Title: Study of Phenotypic and Functional Characteristics of Regulatory T Lymphocytes in Horton's Disease
Acronym: ACG et TREG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SAMSON APJ 2014
Record Dates: First submitted 2016-06-29; First posted 2016-08-05 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Horton's Disease
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Blood Specimen Collection

ARMS (2):
- Horton (Experimental)
  Interventions: Biological: Blood samples
- control (Placebo Comparator)
  Interventions: Biological: Blood samples

INTERVENTIONS:
Biological: Blood samples

SUMMARY:
Giant cell arteritis (GCA) is the most frequent vascularitis after 50 years of age The investigators recently showed that GCA was accompanied by an elevation in Th1 and Th17 response [1]. Even though a quantitative deficit in regulatory TL (Treg) was shown, there are to date no data concerning their precise phenotypic and functional characteristics and notably their ability to inhibit Th1 and Th17 polarisation. The hypothesis of the investigator is that, in GCA, there is quantitative and above all functional deficit of Treg. Recently, progress has been made in the identification of Treg with new markers (CD39), which will make it possible to better identify and to study their specific functions. In this study the phenotypic and functional characteristics of Treg in GCA will be analysed. Better understanding of the role des Treg in GCA should lead to better-targeted treatments for patients with GCA, notably via the blockage of cytokines that inhibit the differentiation and/or function of Treg.

The study is classified interventional because a lot of blood samples are taken.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Patients who have provided written consent
* Patients with national health insurance cover
* Age > 50 years
* Patients with a diagnosis of Horton's disease, before any treatment

Horton's disease is defined by the American College Rheumatology ACR criteria [2], as the association of 3 of the following 5 criteria:

* age at disease onset 50 years or older
* recent onset localized headache
* indurated temporal artery or diminished/abolition of temporal pulse
* erythrocyte sedimentation rate (ESR) greater than 50 mm during the first hour (or C Reactive protein (CRP)>20 mg/L)
* Positive temporal artery biopsy (TAB) showing vascularitis with infiltration by mononuclear cells or granulomatous inflammation with or without giant cells.

Control subjects

Control subjects will be healthy volunteers recruited among blood donors at Dijon University Hospital, voluntary hospital personnel (nurses, doctors, laboratory technicians and secretaries) and patients without infectious, inflammatory or auto-immune diseases or cancer (CRP<5mg/L) recruited in the investigating departments of Dijon Hospital. They will be matched for age and sex and must meet the following criteria:

* Age > 50 years
* Patients with national health insurance cover
* Signed written informed consent form
* Absence of an inflammatory syndrome (CRP<5 mg /L)

Exclusion Criteria:

* Adult under guardianship
* Persons without national health insurance cover
* Pregnant or breast-feeding women
* Patients treated with corticoids or immunosuppressants in the month preceding inclusion
* Patients treated with chemotherapy

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2015-10-05 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Measurement by flow cytometry of the percentage of CD39+ Treg (CD4+CD25highFoxP3+CD39+) among total CD4 TL | through study completion an average of 30 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire, Dijon, France

REFERENCES:
- [Result] Samson M, Greigert H, Ciudad M, Gerard C, Ghesquiere T, Trad M, Corbera-Bellalta M, Genet C, Ouandji S, Cladiere C, Thebault M, Ly KH, Liozon E, Maurier F, Bienvenu B, Terrier B, Guillevin L, Charles P, Quipourt V, Devilliers H, Gabrielle PH, Creuzot-Garcher C, Tarris G, Martin L, Saas P, Audia S, Cid MC, Bonnotte B. Improvement of Treg immune response after treatment with tocilizumab in giant cell arteritis. Clin Transl Immunology. 2021 Sep 12;10(9):e1332. doi: 10.1002/cti2.1332. eCollection 2021. PMID 34532040
- [Derived] Maldiney T, Greigert H, Martin L, Benoit E, Creuzot-Garcher C, Gabrielle PH, Chassot JM, Boccara C, Balvay D, Tavitian B, Clement O, Audia S, Bonnotte B, Samson M. Full-field optical coherence tomography for the diagnosis of giant cell arteritis. PLoS One. 2020 Aug 31;15(8):e0234165. doi: 10.1371/journal.pone.0234165. eCollection 2020. PMID 32866179